CLINICAL TRIAL: NCT01187771
Title: A Randomized Trial of Bariatric Surgery for the Treatment of Sleep Apnea
Brief Title: Apnea, Bariatric Surgery Versus Continuous Positive Airway Pressure (CPAP) Trial
Acronym: ABC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Sanjay R Patel, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HL106410 (NIH); R01HL106410 (NIH)
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic Gastric Banding (Active Comparator)
  Interventions: Procedure: Laparoscopic Gastric Banding
- Continuous Positive Airway Pressure (Active Comparator)
  Interventions: Procedure: Continuous Positive Airway Pressure

INTERVENTIONS:
Procedure: Laparoscopic Gastric Banding — Those randomized to surgery would meet with the bariatric surgeon and the dietitian during the 3 month weight management period and based on insurance requirements, would undergo LGB surgery after 3 months of weight management. PAP therapy would be utilized for the 3 week peri-operative period (1 week prior to 2 weeks post-operatively) given evidence that this might reduce peri-operative respiratory complications. Routine surgical follow-up will occur 2 weeks post-operatively and then every 4-6 weeks to assess weight loss trajectory and adjust the band as needed.
  Arms: Laparoscopic Gastric Banding
Procedure: Continuous Positive Airway Pressure — Participants randomized to the CPAP arm will undergo a CPAP titration within 2 weeks of enrollment unless a split-night study was already performed as part of their diagnostic polysomnogram (PSG) providing a reliable CPAP therapeutic pressure. As soon as an appropriate pressure is identified, CPAP therapy will begin with routinely scheduled follow-up visits to maximize CPAP adherence. All participants will be offered a 12 month supervised weight loss program in addition to OSA-specific therapy.
  Arms: Continuous Positive Airway Pressure

SUMMARY:
The purpose of this study is to assess the feasibility of conducting a comparative effectiveness study comparing a medical versus surgical approach to the initial management of obstructive sleep apnea (OSA) in the setting of obesity.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is one of the most common complications of obesity, resulting in excessive sleepiness and daytime functional impairment as well as acting synergistically with obesity in predisposing to hypertension, insulin resistance, diabetes, cardiovascular disease, and stroke. The current first line treatment for moderate to severe OSA, nasal continuous positive airway pressure (CPAP) is extremely effective but is often not well tolerated, leading to low adherence rates in many patients. Bariatric surgery has been approved as treatment for OSA in patients with co-morbid obesity and in small studies, appears to produce substantial improvements. However, no trials directly comparing bariatric procedures with standard CPAP treatment yet exist to guide clinicians and patients in choosing the most appropriate first line treatment. This trial will address the feasibility and safety, and estimate the effect sizes for a subsequent Phase 3 trial. We will recruit 80 patients with severe OSA and morbid obesity (body mass index, BMI, of 35-45 kg/m2) from two large clinical sleep programs that together care for a wide spectrum and demographically diverse group of OSA patients. After establishing patient and physician equipoise, subjects will be randomized to a trial of CPAP or laparoscopic gastric banding as first line treatment for OSA. The primary outcome measures will be improvement in OSA severity under both ideal and real life conditions (i.e., in the CPAP arm, while using CPAP in a controlled environment vs. while using prescribed therapy in the usual home environment, respectively), which will allow for assessments of both comparative efficacy and effectiveness. Outcomes will be assessed at 9 months to quantify the early effectiveness of each treatment strategy as well as to demonstrate clinical equipoise in conducting a future larger long term trial using these two arms. Further follow-up will occur at 18 months in a subset of 40 patients to determine effect sizes for the subsequent study at a point where the bariatric arm has neared a plateau in weight. Secondary outcomes will include patient-related outcomes including sleepiness, quality of life, and an index of health service utilization. In addition, changes in biomarkers related to inflammation, insulin resistance, lipids, blood pressure, and arterial stiffness will be assessed in each group, and in relationship to changes in BMI and OSA, to identify promising outcome measures for future trials. Incurred costs will be collected in all subjects in order to establish the parameters needed for a cost effectiveness analysis. This pilot study will represent the first controlled comparison of medical and surgical treatments for OSA and in addition, will provide the necessary data to develop the optimal study design for a subsequent long term multi-center comparative effectiveness study to better understand the potential role that bariatric surgery may offer in the management of OSA.

ELIGIBILITY:
Inclusion Criteria:

* Severe sleep apnea with at least 1 referable symptom
* Obesity (BMI 35-45 kg/m2)

Exclusion Criteria:

* Prior use of CPAP within the last two years or prior bariatric surgery
* Hypoxemia or hypercapnia
* Elevated peri-operative risk
* Drowsy driving in past year
* Unstable medical or psychiatric conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay R Patel, M.D., M.S., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

REFERENCES:
- [Result] Dudley KA, Tavakkoli A, Andrews RA, Seiger AN, Bakker JP, Patel SR. Interest in bariatric surgery among obese patients with obstructive sleep apnea. Surg Obes Relat Dis. 2015 Sep-Oct;11(5):1146-51. doi: 10.1016/j.soard.2015.01.006. Epub 2015 Jan 14. PMID 25892349
- [Result] Bakker JP, Tavakkoli A, Rueschman M, Wang W, Andrews R, Malhotra A, Owens RL, Anand A, Dudley KA, Patel SR. Gastric Banding Surgery versus Continuous Positive Airway Pressure for Obstructive Sleep Apnea: A Randomized Controlled Trial. Am J Respir Crit Care Med. 2018 Apr 15;197(8):1080-1083. doi: 10.1164/rccm.201708-1637LE. No abstract available. PMID 29035093

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Between enrollment and assignment, 3 participants withdrew their consent to participate and 1 participant's physician withdrew the determination of eligibility.
Period: Overall Study
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Started | 28 | 21
Completed | 25 | 18
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure | Total
Number analyzed (Participants) | 28 | 21 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 21 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.7 (9.2) | 46.3 (10.5) | 48.8 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 28 | 21 | 49

OUTCOME MEASURES:

1. Primary Outcome: Effective Apnea Hypopnea Index
Description: The Effective Apnea Hypopnea Index (AHI) is the actual frequency of apneas and hypopneas per hour that the patient is exposed to. It is calculated as the AHI while on CPAP times the proportion of sleep time that CPAP was used plus the AHI off CPAP times the proportion of sleep time that CPAP is not used.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Events per hour
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
Events per hour | 29.5 (23.4) | 20.0 (25.3)

2. Primary Outcome: Epworth Sleepiness Score
Description: The Epworth Sleepiness Scale results in scores ranging from 0-24, where scores of 0-10 indicate normal levels of sleepiness while 11-24 indicate excessive daytime sleepiness.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Units on Epworth Sleepiness scale
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
Units on Epworth Sleepiness scale | 7.6 (4.7) | 7.8 (4.8)

3. Secondary Outcome: Mean 24-hour Systolic Blood Pressure
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
mmHg | 121.7 (13.0) | 119.5 (16.8)

4. Secondary Outcome: Insulin Resistance (HOMA Index)
Time Frame: 9 months
Population: Data were not collected.
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Calgary Sleep Apnea Quality of Life Index
Description: The Calgary Sleep Apnea Quality of Life Index results in scores ranging from 1-7, with higher scores indicating a higher quality of life.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: Units on Quality of Life Index
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
Units on Quality of Life Index | 4.8 (0.7) | 4.4 (1.1)

6. Secondary Outcome: Depression (Patient Health Questionnaire-9)
Description: The PHQ-9 is scored from 0-27 with higher scores indicating more severe depression.
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: PHQ-9 scale
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
PHQ-9 scale | 4.0 (3.7) | 6.2 (7.5)

7. Secondary Outcome: Direct Health Care Costs
Time Frame: 9 months
Population: Data not collected.
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Mean 24-hour Diastolic Blood Pressure
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
Number analyzed (Participants) | 25 | 18
mmHg | 75.8 (8.8) | 74.9 (11.0)

ADVERSE EVENTS:
Arm/Group | Laparoscopic Gastric Banding | Continuous Positive Airway Pressure
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/21
Serious Adverse Events (participants affected / at risk) | 5/28 | 2/21
Other Adverse Events (participants affected / at risk) | 25/28 | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laparoscopic Gastric Banding (N=28) | Continuous Positive Airway Pressure (N=21)
Renal disorders (Renal and urinary disorders) | 0 | 1
Urinary tract signs and symptoms (Renal and urinary disorders) | 1 | 0
Anxiety disorders and symptoms (Psychiatric disorders) | 1 | 0
Suicidal and self-injurious behaviors NEC (Psychiatric disorders) | 1 | 1
Gastrointestinal infections (Gastrointestinal disorders) | 1 | 0
Gallbladder disorders (Hepatobiliary disorders) | 1 | 0
Bone and joint injuries (Injury, poisoning and procedural complications) | 0 | 1
Bone disorders (excl congenital and fractures) (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laparoscopic Gastric Banding (N=28) | Continuous Positive Airway Pressure (N=21)
Coronary artery disrders (Cardiac disorders) | 1 | 0
Aural disorders NEC (Ear and labyrinth disorders) | 4 | 2
Ocular infections, irritations and inflammations (Eye disorders) | 1 | 0
Diverticular disorders (Gastrointestinal disorders) | 1 | 1
Gallbladder disorders (Hepatobiliary disorders) | 2 | 0
Gastrointestinal infections (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility (Gastrointestinal disorders) | 1 | 0
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 3 | 2
Dental and gingival conditions (Gastrointestinal disorders) | 0 | 1
Drowsy driving (General disorders) | 6 | 3
Headaches (Nervous system disorders) | 2 | 1
Bone and joint injuries (Injury, poisoning and procedural complications) | 1 | 2
Injuries NEC (Injury, poisoning and procedural complications) | 5 | 4
Medication errors (Injury, poisoning and procedural complications) | 1 | 0
Procedural related injuries and complicatins NEC (Injury, poisoning and procedural complications) | 1 | 0
Glucose metabolism disorders (Metabolism and nutrition disorders) | 1 | 1
Bone disorders (excl congenital and fractures) (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint disorders (Musculoskeletal and connective tissue disorders) | 3 | 3
Muscle disorders (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 1 | 3
Tendon, ligament and cartilage disorders (Musculoskeletal and connective tissue disorders) | 2 | 0
Demyelinating disorders (Nervous system disorders) | 1 | 0
Movement disorders (Nervous system disorders) | 0 | 1
Anxiety disorders and symptoms (Psychiatric disorders) | 0 | 2
Depressed mood disorders and disturbances (Psychiatric disorders) | 1 | 3
Mental impairment disorders (Psychiatric disorders) | 0 | 1
Mood disorders and disturbances NEC (Psychiatric disorders) | 1 | 0
Bladder and bladder neck disorders (excl calculi) (Renal and urinary disorders) | 0 | 1
Genitourinary tract disorders NEC (Renal and urinary disorders) | 1 | 0
Urolithiases (Renal and urinary disorders) | 0 | 2
Female reproductive tract infections and inflammations (Reproductive system and breast disorders) | 2 | 0
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory tract infections (Respiratory, thoracic and mediastinal disorders) | 9 | 9
Upper respiratory tract disorders (excl infections) (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 4 | 0
Skin and subcutaneous tissue infections and infestations (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No